CLINICAL TRIAL: NCT02949180
Title: Enhanced Diagnostics for Early Detection of Atrial Fibrillation - Prospective Validation
Acronym: DETECTAF-pro
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University Hospital Greifswald (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-01176
Record Dates: First submitted 2016-10-27; First posted 2016-10-31 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Atrium; Fibrillation; Arrhythmia Atrial
Keywords: Atrial fibrillation; Rhythm monitoring; Cardiovascular App; m-health
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- AF: Five minutes puls wave recording will be performed in patients in atrial fibrillation at time of recruitment
  Interventions: Device: Five minutes puls wave recording
- SR: Five minutes puls wave recording will be performed in patients in sinus rhythm at time of recruitment
  Interventions: Device: Five minutes puls wave recording

INTERVENTIONS:
Device: Five minutes puls wave recording — iPhone will be positioned on the index finger for five minutes to record a pulse wave

SUMMARY:
Prospective, blinded, multicenter international trial to test the Preventicus Heartbeats App in a prospective cohort.

DETAILED DESCRIPTION:
Introduction This algorithm was validated earlier in a clinical trial with retrospective Data. The results were published accordingly.The algorithm is implemented in the commercial App Preventicus Heartbeats. DETECT AF is designed as prospective follow up trial.

Study design Prospective, blinded, multicenter international trial.

Methods

The subjects will be asked to position a smartphone on their index finger to allow their pulse curve to be recorded for five minutes. At the same time, an ecg will be recorded using an digital mobile ecg recorder as a reference.

Data will be collected on person-related information, comorbidities and medication (estimated overall duration/patient <20 min). No follow-up is planned. Analogous to predecessor studies, the pulse wave curve data are coded with the patient's identification number (ID) and externally analyzed at Preventicus; based on the results, the subjects will be assigned to SR/AF groups. After evaluation of all files, the grouped results will be aggregated, unblinded and evaluated under monitoring.

Primary target parameters are the app's sensitivity and specificity in correctly detecting atrial fibrillation compared to an automatically interpreted ECG.

Secondary target parameters include the proportion of non-evaluable recordings in the overall study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of legal age,
* patients with either sinus rhythm (Group SR) or atrial fibrillation (Group AF)
* informed consent

Exclusion Criteria:

* Legally incompetent persons

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at the University Hospital Basel
Sampling Method: Probability Sample
Enrollment: 672 (Actual)
Dates: Start 2016-10; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Correct detection of atrial fibrillation | 5 minutes
  iPhone will be positioned on the index finger for five minutes to record a pulse wave; Algorithm should correctly differentiate between AF patients and SR patients

CONTACTS AND LOCATIONS:
Overall Officials: Jens Eckstein, MD, PhD, Principal Investigator — Universityhospital Basel
Locations (2):
- University Hospital Greifswald, Greifswald, Germany
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Krivoshei L, Weber S, Burkard T, Maseli A, Brasier N, Kuhne M, Conen D, Huebner T, Seeck A, Eckstein J. Smart detection of atrial fibrillationdagger. Europace. 2017 May 1;19(5):753-757. doi: 10.1093/europace/euw125. PMID 27371660
- [Derived] Brasier N, Raichle CJ, Dorr M, Becke A, Nohturfft V, Weber S, Bulacher F, Salomon L, Noah T, Birkemeyer R, Eckstein J. Detection of atrial fibrillation with a smartphone camera: first prospective, international, two-centre, clinical validation study (DETECT AF PRO). Europace. 2019 Jan 1;21(1):41-47. doi: 10.1093/europace/euy176. PMID 30085018